CLINICAL TRIAL: NCT03703960
Title: Contribution of Hypnotic Analgesia to Local Anesthesia During Bronchial Endoscopy.
Acronym: HypnoFibro
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusion
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GEORGES ADEMPU 2018
Record Dates: First submitted 2018-10-08; First posted 2018-10-12 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Patient With Bronchial Endoscopy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 "Hypnosis" (Experimental)
  Interventions: Other: hypnotic analgesia
- Group 2 "music" (Active Comparator)
  Interventions: Other: music
- Control group (No Intervention)

INTERVENTIONS:
Other: hypnotic analgesia — classic three-step hypnosis procedure (induction, trance and return to consciousness).
  Arms: Group 1 "Hypnosis"
Other: music — calm music conducive to relaxation
  Arms: Group 2 "music"

SUMMARY:
Bronchial endoscopy (or bronchial fibroscopy) is an invasive diagnostic examination performed extremely frequently in the Pneumology department of the Dijon University Hospital, with an average of 1200 procedures per year. It allows the pneumologist to see the first divisions of the bronchial tree but also to take samples for microbiological or anatomopathological purposes. The two main sampling techniques are bronchoalveolar lavage and endobronchial biopsies. Two steps in the process can be unpleasant for the patient:

1. the crossing of the nasopharynx because of the narrow and curving passage,
2. the crossing of the vocal cords and exploration of the trachea, which sometimes causes nausea but especially a cough and a feeling of suffocation.

Depending on the patients, the experience of the examination can be very difficult. In addition, the experience of the examination is influenced by the psychological state of the patient, who is often anxious in the perspective of a diagnosis of a malignancy. It is therefore recommended to perform this examination under local anesthesia (LA) with xylocaine spray 5%. Several protocols, such as the use of atropine, hydroxyzine or benzodiazepines, have been proposed to improve test tolerance, but no pre-medication, other than the drugs indicated in general anesthesia, including midazolam and propofol, has demonstrated their efficacy. Moreover, these molecules are not without respiratory side effects.

Several recent studies have suggested that hypnotic analgesia improves the experience and course of diagnostic procedures that are quite similar to bronchial endoscopy and are usually performed with LA. This is particularly the case for gastroscopy or trans-oesophageal ultrasound. In addition, the effectiveness of hypnotic analgesia for the relief of acute or chronic pain is increasingly well established in the literature. However, the pathophysiology of dyspnea is close to that of pain.

The hypothesis is that adding hypnotic analgesia to the usual local anesthesia will relieve the dyspnea and pain experienced during the examination. There are no studies or data yet on the effect of hypnotic analgesia in bronchial endoscopy with LA. The objective of this work is to demonstrate its effectiveness in order to potentially offer this intervention to all patients and to improve the management of this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given oral consent
* Patient having:

  * a bronchial endoscopy for diagnostic purposes,
  * performed on schedule in the Pneumology Department and Intensive Respiratory Care at the Dijon University Hospital
  * regardless of the indication or samples taken during the examination (simple exploration, lavage, biopsies)

Exclusion Criteria:

* Person not affiliated to a national health insurance system
* Person subject to legal protection (curatorship, guardianship)
* Person under judiciary protection
* Non-menopausal woman
* Adult unable or unwilling to consent
* Minor
* Patient who does not speak French
* Patient with severe hearing disorder that make it difficult to perform hypnosis under good conditions
* Patient with psychiatric or neurological disorders such as dementia, psychosis or profound mental retardation
* Severe COPD requiring long-term oxygen therapy at home or with a tracheotomy
* Patient undergoing bronchial endoscopy for the management of acute respiratory distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
score for the sensory component of dyspnea | through study completion, an average of 30 minutes
  Comparison of the evolution of the score assigned to the sensory component of dyspnea measured by the Multidimensional Dyspnea Profile (MDP) scale before and after bronchial endoscopy between patients of the interventional arm 1 under local anesthesia and hypnotic analgesia, patients of the interventional arm 2 under local anesthesia and relaxing music and patients of the control arm under LA bronchial endoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France